CLINICAL TRIAL: NCT03749902
Title: A Randomized Trial Comparing Oral Misoprostol Alone with Oral Misoprostol Followed by Oxytocin in Women Induced for Hypertension of Pregnancy
Brief Title: A Randomized Trial of Oral Misoprostol Alone Versus Oral Misoprostol Followed by Oxytocin for Labour Induction
Acronym: MOLI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Gynuity Health Projects (Other); Government Medical College, Nagpur (Industry); Daga Memorial Women's Hospital, Nagpur, India (Other); Mahatma Gandhi Institute of Medical Sciences, Sevagram, Wardha, India (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4007
Record Dates: First submitted 2018-11-20; First posted 2018-11-21 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2022-08

CONDITIONS: Induction of Labor
Keywords: preeclampsia; misoprostol; oxytocin
MeSH Terms: conditions — Pre-Eclampsia | interventions — Misoprostol; Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxytocin infusion (Other): * Oxytocin infusion will be given through an electronic infusion pump. One unit of oxytocin will be injected in 500 mL of Ringer's lactate, started at a rate of 2 mU/min, and increased every 30 min by 2 mU/min until there are three to four contractions every 10 min. The rate will be titrated to maintain that contraction frequency. The maximum dose will be 20mU/min as oxytocin summary product characteristics.
  * The oxytocin group will not receive misoprostol after the membranes have ruptured.
  Interventions: Drug: Oxytocin
- Oral misoprostol (Other): * An initial dose of misoprostol 25mcg will be given orally after randomisation (this must be a minimum of 2 hours after the previous misoprostol dose).
  * The next dose of oral misoprostol will be omitted if moderate or strong contractions are occurring at 3 in 10 minutes or more (i.e. 9 or more in the preceding 30 minutes)
  * If contractions subsequently reduce to less than 3 in 10 (under 9 in 30 minutes), or become irregular or mild, then the oral misoprostol 25mcg can be restarted
  * In the event of inadequate progress, clinicians will be advised to give further misoprostol if there are any concerns about contractions strength or frequency.
  Interventions: Drug: Oral misoprostol

INTERVENTIONS:
Drug: Oral misoprostol — * An initial dose of misoprostol 25mcg will be given orally after randomisation (this must be a minimum of 2 hours after the previous misoprostol dose).
  * The next dose of oral misoprostol will be omitted if moderate or strong contractions are occurring at 3 in 10 minutes or more (i.e. 9 or more in the preceding 30 minutes)
  * If contractions subsequently reduce to less than 3 in 10 (under 9 in 30 minutes), or become irregular or mild, then the oral misoprostol 25mcg can be restarted
  * In the event of inadequate progress, clinicians will be advised to give further misoprostol if there are any concerns about contractions strength or frequency.
  Other Names: Misoprost
  Arms: Oral misoprostol
Drug: Oxytocin — * Oxytocin infusion will be given through an electronic infusion pump. One unit of oxytocin will be injected in 500 mL of Ringer's lactate, started at a rate of 2 mU/min, and increased every 30 min by 2 mU/min until there are three to four contractions every 10 min. The rate will be titrated to maintain that contraction frequency. The maximum dose will be 20mU/min as oxytocin summary product characteristics.
  * The oxytocin group will not receive misoprostol after the membranes have ruptured.
  Other Names: Pitocin
  Arms: Oxytocin infusion

SUMMARY:
The primary objective of the trial is to assess the following: In women who have undergone cervical preparation with oral misoprostol as part of labour induction for hypertensive disease in India, is augmentation using oral misoprostol superior to the standard protocol of intravenous oxytocin?

DETAILED DESCRIPTION:
Every year approximately 30 000 women die from hypertensive disease in pregnancy. Magnesium sulphate and anti-hypertensives reduce morbidity, but delivery is the only cure. Low dose oral misoprostol, a prostaglandin E1 analogue, is a highly effective method for labour induction. Usually, once active labour has commenced, the misoprostol is replaced with an intravenous oxytocin infusion. However, some studies have shown that oral misoprostol can be continued into active labour. In the Cochrane review on labour induction, those whose augmentation was continued with misoprostol (M/M protocol) had 42% less CSs than those who changed to oxytocin (M/Ox protocol; 15% vs 26%). This misoprostol-only protocol would be simpler and probably more acceptable to women. However, these two protocols have never been directly compared. We propose a pragmatic, open-label, randomised trial to compare an M/M labour induction protocol with the standard M/Ox protocol.

ELIGIBILITY:
Inclusion Criteria:

* • Ongoing pregnancies with a live fetus who require induction because of preeclampsia or hypertensionWomen will be included irrespective of whether an intrapartum caesarean birth on fetal grounds would be considered or not

  * Women age ≥18 years
  * Signed informed consent form
  * Undergone cervical ripening with misoprostol if cervix initially unfavourable
  * Decision to augment labour for inadequate uterine contractions despite ruptured membranes (either artificial or spontaneous as part of the induction process)s

Exclusion Criteria:

* Women with previous caesarean births
* Those unable to give informed consent
* Cervical ripening with agents other than misoprostol (e.g. Foley catheter, prostaglandins)
* Multiple pregnancy
* History of allergy to misoprostol
* Adequate uterine activity
* Pre- induction Ruptured amniotic membranes
* Frank chorioamnionitis (systemic illness with purulent vaginal discharge and uterine tenderness)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Caesarean birth | At delivery
  Rate of caesarean birth in the treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Weeks, FRCOG, Principal Investigator — University of Liverpool
Locations (3):
- India (3):
  - Daga Memorial Women's Hospital, Nagpur, Maharashtra
  - Mahatma Gandhi Institute of Medical Sciences, Sevāgrām, Maharashtra
  - Government Medical College (GMC), Nagpur

IPD SHARING:
Plan to Share IPD: Yes
The data from this study will be confidential until the database is closed at the end of the study. Following this the study investigators will have exclusive access to the data until the publication of the results in a journal. Once this has happened, the database will be open to other researchers upon request. Open access databases will also be sought so as to maximise the availability of our research data with as few restrictions as possible, in line with MRC and Wellcome Trust policy. The consent form will include a clause for the woman to give permission for her anonymous data to be used for future research studies.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be released upon publication of the trial results. After this, the data will be shared on a public database to maximise the viability of the data.
Access Criteria: Initially this will be upon request with later public publication of the data.

REFERENCES:
- [Derived] Patel A, Howard R, Faragher B, Durocher J, Winikoff B, Symon A, Weeks A, Mundle S, Lightly K. Evaluating women's experiences and satisfaction with labour induction in India: a comparison of the participant generated experience and satisfaction (PaGES) index with standard methods. BMC Pregnancy Childbirth. 2025 May 28;25(1):619. doi: 10.1186/s12884-025-07731-9. PMID 40437451
- [Derived] Symon A, Lightly K, Howard R, Mundle S, Faragher B, Hanley M, Durocher J, Winikoff B, Weeks A. Introducing the participant-generated experience and satisfaction (PaGES) index: a novel, longitudinal mixed-methods evaluation tool. BMC Med Res Methodol. 2023 Sep 28;23(1):214. doi: 10.1186/s12874-023-02016-1. PMID 37759174
- [Derived] Bracken H, Lightly K, Mundle S, Kerr R, Faragher B, Easterling T, Leigh S, Turner M, Alfirevic Z, Winikoff B, Weeks A. Oral Misoprostol alone versus oral misoprostol followed by oxytocin for labour induction in women with hypertension in pregnancy (MOLI): protocol for a randomised controlled trial. BMC Pregnancy Childbirth. 2021 Jul 29;21(1):537. doi: 10.1186/s12884-021-04009-8. PMID 34325670